CLINICAL TRIAL: NCT06936995
Title: Comparison of Preemptive Multimodal Analgesia and Femoral Triangle Block on Early Rehabilitation in ACL Reconstruction: A Prospective, Randomized, Double-Blind Study
Brief Title: Multimodal Analgesia vs. Femoral Block in ACL Surgery
Acronym: MAPvsFTB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, SEVDE NUR AYDIN KUSSAN, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MFT_01
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Injuries; Postoperative Pain; Pain, Postoperative
Keywords: Anterior Cruciate Ligament (ACL) Reconstruction; Postoperative Pain Management; Multimodal Analgesia; Femoral Triangle Block; Rehabilitation Outcomes; Postoperative Recovery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind clinical trial with parallel assignment. Participants will be randomized into two groups to compare the effects of preemptive intravenous multimodal analgesia versus femoral triangle block on early postoperative rehabilitation compliance and pain control following ACL reconstruction surgery.
Who Masked: Participant, Investigator
Masking Description: The study will be double-blind, meaning neither the researchers nor the participants will know which treatment group they belong to, ensuring unbiased outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemptive Multimodal Intravenous Analgesia (Active Comparator): Preemptive multimodal intravenous analgesia protocol, combining opioids, NSAIDs, and adjunctive medications to manage postoperative pain.
  Interventions: Drug: Preemptive Multimodal Intravenous Analgesia
- Femoral Triangle Blok (Experimental): Femoral triangle block, a regional anesthesia technique, to manage postoperative pain by injecting a local anesthetic around the femoral nerve at the femoral triangle point.
  Interventions: Procedure: Femoral Triangle Block

INTERVENTIONS:
Drug: Preemptive Multimodal Intravenous Analgesia — Combination of opioids, NSAIDs, and adjunctive medications to manage postoperative pain before and during surgery.
  Other Names: Multimodal Analgesia; IV Pain Management Protocol
  Arms: Preemptive Multimodal Intravenous Analgesia
Procedure: Femoral Triangle Block — Local anesthetic injection around the femoral nerve to manage postoperative pain via regional anesthesia.
  Other Names: Femoral Nerve Block Anesthesia
  Arms: Femoral Triangle Blok

SUMMARY:
This study aims to compare the effects of a preemptive multimodal intravenous analgesia protocol and a femoral triangle block on early postoperative rehabilitation compliance in patients undergoing anterior cruciate ligament (ACL) reconstruction under general anesthesia. Adult patients aged 18 to 65 will be randomized to receive either multimodal intravenous analgesia or femoral triangle block prior to surgery. Rehabilitation compliance will be evaluated using the straight leg raise test, sit-to-stand success, and pain scores at multiple postoperative time points. Secondary outcomes include opioid consumption, incidence of opioid-related side effects.

DETAILED DESCRIPTION:
Postoperative pain following anterior cruciate ligament (ACL) reconstruction is typically acute in nature and may hinder early physiotherapy interventions. Effective postoperative pain control is essential for optimizing rehabilitation outcomes by enabling early mobilization, which can reduce the risk of thromboembolic complications, maintain pulmonary function, and mitigate metabolic and endocrine stress responses. Adequate analgesia also helps prevent the development of chronic pain, supports cognitive function, and may shorten hospital stay.

ACL injuries are commonly observed in athletes, as well as middle-aged individuals engaging in recreational activities. The success of ACL reconstruction surgery is highly dependent on early and effective postoperative rehabilitation, particularly muscle strength restoration.

Delayed mobilization following surgery may lead to muscle atrophy, cartilage degeneration, and connective tissue adhesions. Early ambulation and rehabilitation are critical for tissue healing and for maintaining joint function and mobility.

Various methods have been utilized for postoperative analgesia, including patient-controlled epidural analgesia, intravenous patient-controlled analgesia (PCA), peripheral nerve blocks, and intra-articular local anesthetic infiltration. Multimodal analgesia protocols have demonstrated superior outcomes in terms of pain control, opioid-sparing effects, and patient satisfaction when compared with single-modality approaches.

This prospective, randomized, double-blind clinical trial will compare the effects of preemptive intravenous multimodal analgesia and femoral triangle block on early postoperative rehabilitation compliance in adult patients undergoing ACL reconstruction under general anesthesia. The interventions are routinely used in clinical practice and are recognized as safe and effective.

The primary objective is to evaluate whether either approach improves compliance with early rehabilitation tasks. Compliance will be assessed using functional recovery metrics including the straight leg raise test, sit-to-stand success, and patient-reported pain scores using the Numerical Rating Scale (NRS) at predefined postoperative time points.

Secondary endpoints include total opioid consumption, frequency of opioid-related adverse events (e.g., nausea, vomiting, itching), and overall patient satisfaction. This study addresses a current gap in the literature, as no previous trials have directly compared these two methods in this clinical context.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 years or older. Condition: Patients scheduled for anterior cruciate ligament (ACL) reconstruction surgery.

ASA Classification: Patients classified as ASA I, II, or III. Orientation: Patients who are fully oriented and can cooperate with study procedures.

Consent: Patients capable of providing informed consent to participate in the study.

Exclusion Criteria:

Informed Consent: Patients unable to provide informed consent. BMI: Patients with a BMI of ≥30 kg/m². Allergy: Known allergy to local anesthetics. Orientation and Cooperation: Patients who are not fully oriented or cannot cooperate with study procedures.

Additional Trauma: Patients with other traumatic injuries requiring opioid analgesia.

Neuropathic Pain History: Patients with a history of neuropathic pain. Chronic Pain Syndrome: Patients with a history of chronic pain syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Compliance with Straight Leg Raise Test (SLR) | Postoperative 2, 6, 12 and 24 hours
  This outcome measure evaluates the patients' ability to perform the straight leg raise test (SLR) at various postoperative time points. The NRS (Numeric Rating Scale) score will be used to assess the pain during these activities. NRS (Numeric Rating Scale) for pain during the activity. Scale: 0 (no pain) to 10 (worst pain). Higher scores on the NRS indicate worse pain.
Standing Ability | Postoperative 2,6,12 and 24 hours
  This outcome measure evaluates the patients' ability to stand after surgery at various postoperative time points. The NRS (Numeric Rating Scale) score will be used to assess the pain during these activities. NRS (Numeric Rating Scale) for pain during the activity. Scale: 0 (no pain) to 10 (worst pain). Higher scores on the NRS indicate worse pain.

SECONDARY OUTCOMES:
Total Opioid Consumption | Postoperative 2, 6, 12, 24, 48, and 72 hours
  The total amount of opioids consumed by the patients in the first 72 hours after surgery will be recorded and compared between the two groups.
Incidence of Opioid-Related Side Effects | Postoperative 2, 6, 12, 24, 48, and 72 hours
  The incidence of opioid-related side effects, such as nausea, vomiting, and itching, will be recorded and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: MENEKŞE ÖZÇELİK, Study Director — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No